CLINICAL TRIAL: NCT05165303
Title: Minimal Effective Concentration of Lidocaine in Propofol Lidocaine Mixture for Relief of Pain on Propofol Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hitham Mohammed Aly Elsayed, Anesthesia consultant, Imam Abdulrahman Bin Faisal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-331-KFUH
Record Dates: First submitted 2021-10-16; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Propofol

STUDY DESIGN:
Intervention Model Description: clinical trial with a single arm
Masking Description: Mixtures of propofol, lidocaine and saline will be prepared by an anesthetist who is not involved in the study team, participants, investigator and anesthesia care giver will be blinded for the lidocaine concentration used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lidocaine with propofol (Experimental)
  Interventions: Drug: lidocaine with propofol

INTERVENTIONS:
Drug: lidocaine with propofol — different concentrations of lidocaine added to propofol varying from

SUMMARY:
The research will be carried out in order to determine the optimal lidocaine concentration in propofol lidocaine mixture to prevent pain on propofol injection during induction of general anesthesia using a modified Dixon's up-and-down method. We hypothesized that focusing on lidocaine concentration and not dose could be more convenient and valuable to alleviate pain with propofol injection.

Patients & methods include assessment of severity of pain on propofol injection using nine concentrations of lidocaine in lidocaine propofol mixture in ASA I&II patients aged 16-60 years with excluxion of patients with history of drug allergy, hepatic or renal impairment, cardiac problems, neurologic deficits or psychiatric disorders.

Demographic data, type and duration of surgery, Time for unconsciousness, volume of propofol-lidocaine mixture used, pain scale during injection, increase in heart rate and/or hand or forearm withdrawal during injection will be recorded and patient satisfaction (will be assessed in the recovery room after regaining consciousness),

DETAILED DESCRIPTION:
The research will be carried out in order to determine the optimal lidocaine concentration in propofol lidocaine mixture to prevent pain on propofol injection during induction of general anesthesia using a modified Dixon's up-and-down method. We hypothesized that focusing on lidocaine concentration and not dose could be more convenient and valuable to alleviate pain with propofol injection.

Patients & methods include assessment of severity of pain on propofol injection using nine concentrations of lidocaine in in lidocaine propofol mixture in ASA I&II patients aged 18-60 years with exclusion of patients with history of drug allergy, hepatic or renal impairment, cardiac problems, neurologic deficits or psychiatric disorders.

Demographic data, type and duration of surgery, Time for unconsciousness, volume of propofol-lidocaine mixture used, pain scale during injection, increase in heart rate and/or hand or forearm withdrawal during injection, patient satisfaction (will be assessed in the recovery room after regaining consciousness),

ELIGIBILITY:
Inclusion Criteria:

* ASA I &II
* Age 18 - 60 years

Exclusion Criteria:

* study drug allergy
* hepatic or renal impairment
* cardiac problem
* neurologic deficits
* psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
propofol injection pain | during injection untill patient start loosing conciousness
  burning pain felt by the participant during injection of propofol according to pain scale including mild, moderate and severe pain degrees

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mohammed, MD, Study Director — King Fahd university hospital

IPD SHARING:
Plan to Share IPD: No